CLINICAL TRIAL: NCT01520558
Title: A Phase 1/2 Study of CNDO-109-Activated Allogeneic Natural Killer Cells in Patients With High Risk Acute Myeloid Leukemia in First Complete Remission (CR1)
Brief Title: CNDO-109-AANK for AML in First Complete Remission (CR1)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coronado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNDO109-001
Record Dates: First submitted 2012-01-24; First posted 2012-01-30 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; High Risk Relapse; Complete Remission; Allogeneic Natural Killer Cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CNDO-109-AANK Cells Dose 1 (Experimental): In stage 1, patients will receive one of three doses of CNDO-109-AANK cells, and the lowest of these three doses (dose 1) is 3×10^5 cells/kg recipient body weight. In stage 2, the MTD will have been determined and all patients will receive either Dose 1, Dose 2 or Dose 3.
  Interventions: Biological: CNDO-109-AANK Cells
- CNDO-109-AANK Cells Dose 2 (Experimental): In stage 1, patients will receive one of three doses of CNDO-109-AANK cells, and the middle dose of these three doses (dose 2) is 1×10^6 cells/kg recipient body weight. In stage 2, the MTD will have been determined and all patients will receive either Dose 1, Dose 2 or Dose 3.
  Interventions: Biological: CNDO-109-AANK Cells
- CNDO-109-AANK Cells Dose 3 (Experimental): In stage 1, patients will receive one of three doses of CNDO-109-AANK cells, and the highest dose of these three doses (dose 3) is 3×10^6 cells/kg recipient body weight. In stage 2, the MTD will have been determined and all patients will receive either Dose 1, Dose 2 or Dose 3.
  Interventions: Biological: CNDO-109-AANK Cells

INTERVENTIONS:
Biological: CNDO-109-AANK Cells — Single dose, infusion
  Other Names: CNDO-109-Activated Allogeneic Natural Killer Cells

SUMMARY:
This is a multi-center, open-label, non-controlled, non-randomized dose-escalating Phase 1 clinical study designed to examine the safety of infusing escalating doses of CNDO-109-Activated Allogeneic Natural Killer Cells-(from a first or second degree relative), after a preparatory chemotherapy regimen, in adult patients with acute myeloid leukemia (AML) who are in their first complete remission at the time of enrollment, are not candidates for stem cell transplant, and are considered to be at high risk for recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has pathologically documented AML and is in CR1 at the time of the screening visit
2. The patient achieved CR1 within 10 weeks of the screening visit; the patient may have received post-remission consolidation therapy (except for transplant) prior to the screening visit
3. A bone marrow aspiration performed within 21 days prior to the start of pre-infusion preparative therapy confirms the patient is in CR1
4. The patient has either refused or is not considered an appropriate immediate candidate for transplantation and is considered to be at high risk for recurrence by having at least one of the following prognostic factors:

   * High risk cytogenetics (-5, -7, del(5q), abnormal 3q, 11q23 translocations, complex cytogenetics) or if cytogenetics are normal the presence of a FLT3 mutation without a NPM1 mutation
   * Age > 60 years
   * Antecedent hematological disorder (AHD)
   * AML that is considered to be therapy-related
   * FAB subtype M0 (minimally differentiated acute myeloblastic leukemia), M6 (acute erythroid leukemias, including erythroleukemia (M6a) and pure erythroid leukemia (M6b)), or M7 (acute megakaryoblastic leukemia)
5. The patient is male or female, age 18 years or older
6. The patient has an ECOG performance status of 0, 1, or 2
7. The patient has an available NK cell donor who is a HLA haploidentical first-degree (parent, child, or sibling) or second-degree (child of a sibling) relative; minimum testing will be for HLA-A, HLA-B, and HLA-DR with donors matched for 3/6, 4/6 or 5/6 antigens
8. The patient has an absence of coexisting medical problems that would significantly increase the risk of the chemotherapy procedure (e.g. poor left ventricular ejection fraction [LVEF<40%])
9. The patient has recovered from reversible toxicity from prior therapy. Permanent and stable side effects or changes are acceptable if ≤ Grade 1 (CTCAE, v4.03)
10. The patient has serum creatinine <2×ULN and not rising for at least 2-4 weeks before chemotherapy. If elevated, the 24-hour creatinine clearance must be >50 mL/min
11. The patient has serum total bilirubin < 2 g/dL (unless the patient has a diagnosis of Gilbert's disease), SGOT (ALT) <3.5×ULN, and SGPT (AST) <3.5×ULN
12. The patient has an absolute neutrophil count (ANC) ≥1000/µL, platelets ≥100,000/µL and is not transfusion dependent for platelets and/or red cells
13. The patient has LVEF ≥40% by ECHO or MUGA scan and no clinically significant abnormalities in 12-lead ECG
14. The patient has a PT (or INR) and PTT up to 1.25×ULN
15. The patient must not be dependent on supplemental oxygen
16. The patient is using an effective contraceptive (per the institutional standard), if procreative potential exists
17. The patient must be willing and able to comply with all study protocol requirements. The patient or a legally authorized representative must fully understand all elements of the informed consent and have signed the informed consent according to institutional and federal regulatory requirements
18. The patient has not received an investigational chemotherapy within the last 28 days prior to the screening visit and has never received investigational immunotherapy. In addition, the patient must not receive treatment for AML (including treatment with IL-2 or IFNγ) in the interval of time between the screening visit and initiation of pre-infusion preparative therapy

Exclusion Criteria:

1. The patient had a previous bone marrow or stem cell transplant
2. The patient is seropositive for HIV 1, HIV 2, HBV, or HCV
3. The patient has a psychiatric, addictive, neurological or other disorder that compromises the ability to give informed consent or comply with study requirements
4. The patient is pregnant (confirmed by urine or serum pregnancy test) or lactating
5. The patient has a recently diagnosed active malignancy requiring therapy
6. The patient has an uncontrolled infection, or is receiving anti-fungal treatment for an ongoing infection
7. The patient has known hypersensitivity to bovine proteins
8. The patient has any condition that will place the patient at undue risk or discomfort as a result of adherence to study procedures
9. The patient requires treatment with corticosteroids at a dose > 0.1 mg/kg/day or has a known allergy to DSMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Actual); Study Completion 2018-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Minnesota - Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CNDO-109-AANK Cells Dose 1 | CNDO-109-AANK Cells Dose 2 | CNDO-109-AANK Cells Dose 3
Started | 3 | 3 | 6
Completed | 1 | 1 | 3
Not Completed | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CNDO-109-AANK Cells Dose 1 | CNDO-109-AANK Cells Dose 2 | CNDO-109-AANK Cells Dose 3 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (1.00) | 76.3 (2.52) | 67.3 (6.35) | 71.0 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 4
  Male | 0 | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Define MTD
Description: The primary objective is to define the maximum tolerated dose (MTD), or the maximum tested dose where multiple dose-limiting toxicities (DLTs) are not observed, of CNDO-109-Activated Allogeneic Natural Killer Cells infused after preparative chemotherapy, administered to patients with acute myeloid leukemia (AML) who are in their first complete remission (CR1) at the time of enrollment and are considered to be at high risk for recurrence. The MTD outcome measure is presented as number of participants with DLTs.
Time Frame: up to 30 days post dose
Measure: Count of Participants; unit: Participants
Arm/Group | CNDO-109-AANK Cells Dose 1 | CNDO-109-AANK Cells Dose 2 | CNDO-109-AANK Cells Dose 3
Number analyzed (Participants) | 3 | 3 | 6
Participants | 3 | 3 | 6

2. Secondary Outcome: Additional Safety Profile Beyond MTD
Description: Characterize the safety profile of CNDO-109-Activated Allogeneic Natural Killer Cells infusion after preparative therapy by measurement of adverse events, safety labs, vital signs, bone marrow biopsy/aspiration and physical examination.
Time Frame: up to 360 days post dose
Reporting Status: Not Posted

3. Secondary Outcome: Efficacy
Description: Determine relapse free survival (RFS) and overall survival (OS) following infusion with CNDO-109-Activated Allogeneic Natural Killer Cells.
Time Frame: from the date of documented CR until the first documented progression date or until day 360 post dose whichever is sooner
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | CNDO-109-AANK Cells Dose 1 | CNDO-109-AANK Cells Dose 2 | CNDO-109-AANK Cells Dose 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNDO-109-AANK Cells Dose 1 (N=3) | CNDO-109-AANK Cells Dose 2 (N=3) | CNDO-109-AANK Cells Dose 3 (N=6)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNDO-109-AANK Cells Dose 1 (N=3) | CNDO-109-AANK Cells Dose 2 (N=3) | CNDO-109-AANK Cells Dose 3 (N=6)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
WBC count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Lymph count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
ALT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Alk Phos increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymph count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperurecemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement is specific to clinical trial agreement